CLINICAL TRIAL: NCT07123181
Title: Effects of Increasing Polyphenol Intake by Consumption of Oregano and Basil Leaves on Plasma Inflammatory and Lipid Factors and Total Urinary Polyphenol in Patients With Unstable Angina
Brief Title: Oregano and Basil Leaves and Coronary Artery Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Javad Nasrollahzadeh, Associate Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 43010795
Record Dates: First submitted 2025-08-08; First posted 2025-08-14 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-08

CONDITIONS: Acute Coronary Syndromes; Unstable Angina (UA)
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Standard medical treatment
  Interventions: Other: Control (Standard treatment)
- Higher polyphenol intake by consumption of oregano and basil (Experimental): Daily consumption of oregano and basil leaves along with standard medical treatment
  Interventions: Other: Higher polyphenol intake by consumption of oregano and basil

INTERVENTIONS:
Other: Control (Standard treatment) — Patients receive standard medical treatment.
  Arms: Control
Other: Higher polyphenol intake by consumption of oregano and basil — Patients consume 4-5 grams of dried oregano and 4-5 grams of dried basil leaves daily for two months in addition to their usual medical treatment.
  Arms: Higher polyphenol intake by consumption of oregano and basil

SUMMARY:
The present study will examine the effects of increasing dietary polyphenol intake by consumption of oregano and basil leaves, on plasma inflammatory and lipid factors and total urinary polyphenol levels in patients who have recently had unstable angina.

DETAILED DESCRIPTION:
Several epidemiological studies have shown an inverse relationship between polyphenol consumption and the incidence of chronic diseases, including cardiovascular disease. Dietary polyphenols can act as antioxidants, neutralizing free radicals and reactive oxygen species produced during inflammation. This can helps prevent cellular damage and alleviate oxidative stress-related inflammation. In order to increase the intake of dietary polyphenols, the consumption of vegetables and whole grains has been emphasized, along with the average amount of fruit, fungi, and algae. Moreover, it has been reported that a wider diversity of intake of polyphenols and flavonoid-rich foods when consumed together may represent the optimal approach for improving long-term health. Oregano and basil leaves are two aromatic herbs that are frequently utilized as flavorings in culinary preparations. However, in certain culinary traditions, these herbs are also consumed as part of the daily diet in the form of leafy greens. These herbs have been demonstrated to be excellent sources of polyphenols, particularly rosmarinic acid. The ingestion of these herbs has been shown to augment the dietary intake of beneficial phytochemicals and to support overall antioxidant status. . In addition, these herbs contain active compounds with potential capacity to modulate plasma lipid levels in a beneficial manner that can contribute to the protection of cardiovascular health.

Given the high content of polyphenols in basil and oregano leaves and their potential properties in reducing inflammation and modulating lipids, their consumption may help reduce risk factors associated with coronary heart disease, including unstable angina. The present study will examine the effects of increasing dietary polyphenol intake by consumption of oregano and basil leaves, on plasma inflammatory and lipid factors and total urinary polyphenol levels in patients who have recently had unstable angina.

The present study utilizes a randomized controlled clinical trial design. In this study, patients who meet the established eligibility criteria and are referred to Imam Husain hospital will be included in the study sample. Patients will be randomly assigned to one of two study groups: the control group and the herbs group. The study is scheduled to be conducted over the course of two months. The control group will receive standard medical treatment and general dietary advice, including recommendations to reduce salt, fat, and simple sugar intake. In the herbs group, in addition to the aforementioned recommendations, patients will consume 4-5 grams of dried basil leaves and 4-5 grams of oregano leaves per day. All patients will avoid taking any over-the-counter herbal medications or dietary supplements during the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with unstable angina

Exclusion Criteria:

* Patients diagnosed with STEMI
* Patients undergoing coronary artery bypass grafting
* Liver cirrhosis and advanced chronic kidney disease (CKD 5)
* Having known inflammatory and autoimmune diseases, such as inflammatory bowel disease (IBD) and rheumatoid arthritis, or taking glucocorticoid medications
* Pregnancy or breastfeeding

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-17 (Estimated); Study Completion 2026-06-02 (Estimated)

PRIMARY OUTCOMES:
Plasma inflammatory biomarkers | At the beginning of the study and two months later
  Plasma c-reactive protein, Interleukin-6, RANTES (CCL5)
Plasma lipids | At the beginning of the study and two months later
  Plasma concentrations of triglyceride, cholesterol, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol

SECONDARY OUTCOMES:
Plasma malondialdehyde | At the beginning of the study and two months later
  Plasma concentrations of malondialdehyde
Urinary total polyphenols | At the beginning of the study and two months later
  Levels total polyphenols in spot urine sample measured by Folin-Ciocalteu method
Plasma PCSK9 and PAI-1 levels | At the beginning of the study and two months later
  plasma concentrations of proprotein convertase subtilisin/kexin type 9 (PCSK9) and plasminogen activator inhibitor 1 (PAI-1)

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Husain hospital, Tehran, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided